CLINICAL TRIAL: NCT05172804
Title: The Distinct Effects of Mind-Body Modalities on Health Outcomes in Nursing Students
Brief Title: Mind-Body Modalities for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5/121/2019
Record Dates: First submitted 2021-11-24; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Stress Reaction; Stress, Psychological; Stress, Physiological
Keywords: Stress; Students; Nursing; Mind-body modalities; Mindfulness meditation; Progressive muscle relaxation; Guided imagery; Health outcomes
MeSH Terms: conditions — Fractures, Stress; Stress, Psychological | interventions — Autogenic Training; Imagery, Psychotherapy; Mindfulness; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nursing students receiving progressive muscle relaxation (Experimental): PMR (Smith Version) involves a tense-let go exercise of 11 muscle groups including hand, arm, arm and sides, back, shoulder, face, front of neck, stomach, chest, leg, and foot. This tense-let go exercise is performed twice for each muscle group. The tensing up phase for each muscle group should last for 5 to 10 seconds and the letting go phase for 20-30 seconds. Simultaneously, the subjects will be asked to pay attention to the sensations of muscle tension and relaxation. After the tense-let go exercise, subjects are asked to systematically scan the muscle groups to notice and let go any remaining muscle tension. The entire exercise should take around 30 minutes, not counting instructions and times of measurement [11].
  Interventions: Behavioral: Progressive muscle relaxation
- Nursing students receiving guided imagery (Experimental): Guided imagery (Smith Version) involves creating in one's mind or imagining a passive relaxing places or activities. In sense imagery, one simply imagines sensations associated with a relaxing setting or activity. The relaxation approach involves the sense of sight, sound, touch, and smell. The categories of stimuli consist of: (1) Travel such as boats, plains, trains, balloons, horses, (2) outdoor nature settings such as mountains, gardens, and forest, (3) water such as rivers, lakes, ocean, beach, rain, and (4) indoor settings such as childhood home, castle, religious institution, and cabin [11].
  Interventions: Behavioral: Guided Imagery
- Nursing student receiving mindfulness meditation (Experimental): Smith version of the mindfulness meditation will be used in the current study. The mindful mediators are neutral observers who view the world as it is, without reactions, judgments, and evaluations. They quietly attend to, note, and let go of every internal external stimulus such as thought, feeing, sensation, sound, idea that enters awareness. They do not try to think about, push away, and do anything with these stimuli experienced and do not have to figure out the connections between each stimulus. They simply let each stimulus come and go and wait for the next stimulus. They do not have to be concerned about distractions. Each time they are distracted, they note it as yet another passing stimulus (Ah, a distraction… how interesting") [11].
  Interventions: Behavioral: Mindfulness Meditation
- control Group (Active Comparator): Participants in the control condition will be instructed to sit with their eyes closed during the intervention periods. Participants in the control group will follow an identical time periods as the experimental groups. For instance, when the experimental groups will practice for 30 minutes, the participants in the control group will be asked to sit with eyes closed and relax for 30 minutes.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Progressive muscle relaxation — PMR (Smith Version) involves a tense-let go exercise of 11 muscle groups including hand, arm, arm and sides, back, shoulder, face, front of neck, stomach, chest, leg, and foot. This tense-let go exercise is performed twice for each muscle group. The tensing up phase for each muscle group should last for 5 to 10 seconds and the letting go phase for 20-30 seconds. Simultaneously, the subjects will be asked to pay attention to the sensations of muscle tension and relaxation. After the tense-let go exercise, subjects are asked to systematically scan the muscle groups to notice and let go any remaining muscle tension. The entire exercise should take around 30 minutes, not counting instructions and times of measurement [11].
  Arms: Nursing students receiving progressive muscle relaxation
Behavioral: Guided Imagery — Guided imagery (Smith Version) involves creating in one's mind or imagining a passive relaxing places or activities. In sense imagery, one simply imagines sensations associated with a relaxing setting or activity. The relaxation approach involves the sense of sight, sound, touch, and smell. The categories of stimuli consist of: (1) Travel such as boats, plains, trains, balloons, horses, (2) outdoor nature settings such as mountains, gardens, and forest, (3) water such as rivers, lakes, ocean, beach, rain, and (4) indoor settings such as childhood home, castle, religious institution, and cabin [11].
  Arms: Nursing students receiving guided imagery
Behavioral: Mindfulness Meditation — Smith version of the mindfulness meditation will be used in the current study. The mindful mediators are neutral observers who view the world as it is, without reactions, judgments, and evaluations. They quietly attend to, note, and let go of every internal external stimulus such as thought, feeing, sensation, sound, idea that enters awareness. They do not try to think about, push away, and do anything with these stimuli experienced and do not have to figure out the connections between each stimulus. They simply let each stimulus come and go and wait for the next stimulus. They do not have to be concerned about distractions. Each time they are distracted, they note it as yet another passing stimulus (Ah, a distraction… how interesting") [11].
  Arms: Nursing student receiving mindfulness meditation
Other: Control group — Participants in the control condition will be instructed to sit with their eyes closed and relax during the intervention periods. Participants in the control group will follow an identical procedure and time periods as the experimental groups. For instance, when the experimental groups will practice for 30 minutes, the participants in the control group will be asked to sit with eyes closed and relax for 30 minutes.
  Arms: control Group

SUMMARY:
Background: Nursing students around the world can experience tremendous stress due to their multi-faceted responsibilities. Stress is related to negative health and academic outcomes. Mind-body connection modalities have been used successfully to reduce stress and improve health among healthy and ill individuals in various cultures, but their effects have not yet been studied in the Arab culture. Thus, the purpose of this study was to examine and compare the effects of three of such modalities including progressive muscle relaxation (PMR), guided imagery (GI), and mindfulness meditation (MM) on stress and health outcomes in Jordanian nursing students.

Methods: Using a randomized controlled design, 124 nursing students will be randomly assigned to 4 groups at a large university in Jordan. The 3 experimental groups (PMR, GI, and MM) will participate in 5 30-minute sessions (one session/week for 5 weeks) led by experienced trainers, in a private room during their clinical days. The control group will stay calm for 30 minutes during introducing the study interventions in another room at the university. The health outcomes will be measured at baseline (Time 1) and the end (Time 3) of the intervention in each group using different physical and self-report measures classified into different health categories such as cognitive health outcomes (executive brain function, stressful appraisal, mindfulness), physical health outcomes (e.g. physical symptoms, heart rate, blood pressure, neurobiological markers such as dopamine, serotonin, cortisol, adrenaline, and noradrenaline), and psychological health outcomes (e.g. depression, anxiety).

DETAILED DESCRIPTION:
Design

This study uses a blocked randomized controlled design. The study subjects will be selected using a convenience sampling method. When selected, the subjects will be randomly assigned to either one of the 4 study groups using a stratified random strategy (stratifying variable= academic year of study). The study groups (PMR, MM, GI, Control group) will received 5 30-minute weekly sessions of their assigned intervention over 5 weeks. However, there will be a 4-hours workshop explaining the purposes and techniques of the study interventions before introducing the actual session. The subjects will be asked and encouraged to practice their assigned intervention for 30 minutes daily at home. The dependent variables will be measured three times for the 4 groups: at baseline, at the middle (after the second session), and at the end of intervention.

Participants

Participants are undergraduate nursing students who will be selected using a random sampling method from Jordan University of Science and Technology.

Determination of Sample Size

Using G* Power software 3.1, mixed-design (within groups-between groups) repeated measures ANOVA, an alpha of .05, a power of 0.8, the number of measurements of 3, the number of groups of 4, and a moderate effect size of 0.25, the sample size of 180 was generated. A 15 % attrition rate was reported in a previous study with variables similar to the present study. Considering an expected attrition rate of 15 %, the required final total sample size 210.

Intervention

In the current study, the Attentional Behavioral Cognitive (ABC) Relaxation theory's standardized versions of PMR, MM, and GI will be used, including 5 30-minute weekly sessions of each version. Each group will be encouraged to practice once at home daily. An additional educational 4-hour workshop about each intervention will be provided before the actual training session to enhance the subjects' understanding of their assigned intervention. Especially such interventions are rarely practiced and little known about them in Jordan. In the initial educational session, the PI will separately provide a power point presentation to participants in each experimental group about the rationale and procedures of their assigned intervention and a demonstration of the entire intervention protocol. Participants will be asked briefly to practice their assigned intervention and then evaluated by the PI to make sure the interventions have been done correctly. The PI will give the participants the opportunity to ask questions during the educational session During the actual training sessions, the interventions will be introduced to subjects in the experimental groups using an audio drive designed and produced by the PI based on the ABC Relaxation Theory's guidelines and protocols. All groups will be given identical instructions; only the specific instructions regarding the intervention will be different. The participants in all groups will be asked to close their eyes. All of the groups will be meet in an academic classroom, where the interventions will be provided. Participants will sit in hard chairs behind a desk. Floors will be hard tile. Lights will be dimmed during relaxation phases, and turned on when measures will be filled out. The study groups will be given a audio drive about their assigned intervention and encouraged to practice their assigned intervention daily over the study. They will be asked to document their practices of the assigned intervention at home. The PI will randomly select sessions to evaluate the delivery of intervention using checklists produced according to the developed protocols. PI is an experienced practitioner who received a stress management training at the Psychology Department, Kent State University 7 years ago. Since then, PI has been practicing the stress management techniques daily, especially used in the current study.

Progressive Muscle Relaxation

PMR (ABC Relaxation Theory Version) involves a tense-let go exercise of 11 muscle groups including hand, arm, arm and sides, back, shoulder, face, front of neck, stomach, chest, leg, and foot. This tense-let go exercise is performed twice for each muscle group. The tensing up phase for each muscle group should last for 5 to 10 seconds and the letting go phase for 20-30 seconds. Simultaneously, the subjects will be asked to pay attention to the sensations of muscle tension and relaxation. After the tense-let go exercise, subjects are asked to systematically scan the muscle groups to notice and let go any remaining muscle tension. The entire exercise should take around 30 minutes, not counting instructions and times of measurement.

Guided Imagery

Guided imagery (ABC Relaxation Theory Version) involves creating in one's mind or imagining a passive relaxing places or activities. In sense imagery, one simply imagines sensations associated with a relaxing setting or activity. The relaxation approach involves the sense of sight, sound, touch, and smell. The categories of stimuli consist of: (1) Travel such as boats, plains, trains, balloons, horses, (2) outdoor nature settings such as mountains, gardens, and forest, (3) water such as rivers, lakes, ocean, beach, rain, and (4) indoor settings such as childhood home, castle, religious institution, and cabin.

Mindfulness Meditation

The ABC Relaxation Theory Version of the mindfulness meditation will be used in the current study. The mindful mediators are neutral observers who view the world as it is, without reactions, judgments, and evaluations. They quietly attend to, note, and let go of every internal external stimulus such as thought, feeing, sensation, sound, idea that enters awareness. They do not try to think about, push away, and do anything with these stimuli experienced and do not have to figure out the connections between each stimulus. They simply let each stimulus come and go and wait for the next stimulus. They do not have to be concerned about distractions. Each time they are distracted, they note it as yet another passing stimulus (Ah, a distraction… how interesting").

Control Group

Participants in the control condition will be instructed to sit with their eyes closed and relax during the intervention periods. Participants in the control group will follow an identical procedure and time periods as the experimental groups. For instance, when the experimental groups will practice for 30 minutes, the participants in the control group will be asked to sit with eyes closed and relax for 30 minutes.

Procedure

First, approvals from the JUST institutional review boards will be obtained. After that, a translation from English to Arabic and pilot testing of the English versions of the scales used in the current study will be performed. The scales used in the study will be introduced for 30 Jordanian undergraduate nursing students, and then the construct validity, reliability (internal consistency), readability of these scales will be examined.

After taking the permission of the dean of nursing college and class's instructors, the PI will visit students in their classrooms. As the lecture finishes, The PI will make an announcement about the title and objectives of the study and ask the students who would like to participate to contact him using a business card including the PI's contact information (his name, phone number, and email) given for each one. The contact information will be used only for the purpose of the study. The PI will arrange an initial meeting to meet with students who would like to participate on another day in a private room at the university. At this meeting, the PI will inform the students the study's objectives, risks, benefits, and confidentiality and answer questions that they have about the study. Also, they will be assured that they have the full right to refuse or discontinue the participation at any time and that such refusal or discontinuation will not affect their academic achievements in any way. If agree to participate and eligibility criteria are met, informed consent will be obtained at the meeting. After that, the participants will be randomly assigned equally to the study groups using a stratified random assignment method (stratifying variable= academic year of study). Finally, dates and times for sessions will be set up and sent to the participants using their e-mails.

In the 4-hour education session, the baseline measurements of the study variables will first be obtained. Then the PI will separately provide a power point presentation to participants in each experimental group as explained previously. At the end of the workshop, to avoid experiment contamination, the participants in each experimental group will be asked not to share any information related to the intervention with subjects in other groups.

The actual training will be introduced to subjects in the experimental groups, using an audio CD designed and produced by the PI based on the interventions' guidelines and protocols. Based on the ABC Relaxation Theory (Smith, 2005), at least two, and preferably five sessions of actual mind-body training should be provided to evoke relaxation and optimize health. In the proposed study, the dependent variables will be measured at the middle and at the end of intervention to see whether further health benefits occur between these two measurements. The sessions will be provided to the study groups in a private, quiet, comfortable, and spacious room at the university. The dependent variables will be measured three times for the groups: at baseline, after 2nd actual training session, and at the end of intervention (after 5th session), as mentioned previously.

Various strategies will be followed to decrease measurement errors potentially affected by variations of data collection procedure. For example, filling out the questionnaire may be stressful for some subjects and, in turn, influences objective measures. Therefore, the self-reports measures will be completed after taking the objective measures. Also, all study measurements in the intervention and control groups will be undertaken in the same conditions (i.e. same room temperature and environment) by well-trained nurses as much as possible. The ELISA protocol, including blood sampling will strictly be followed. The neurotransmitters/hormones will measured between 8:30 and 9:30 am for all subjects at sitting position. Drinking coffee, tea, and having should be avoided 6 hours before the measurement of neurotransmitters/hormones. To decrease venipuncture-related pain during blood sampling, EMLA cream will be used, which has been found effective in decreasing venipuncture-related pain in different populations. In addition, quiet environments, free from distraction, will be maintained with a "Do Not Disturb" sign on the door of the rooms during the intervention and data collection.

Statistical Analysis

Statistical analysis will be conducted using SPSS software (version 23). Descriptive statistics will be used to describe the sample. The sample and variables will be described by measures of central tendency and dispersion appropriate to the level of measurement. Initial analyses will be conducted to ensure that the randomization across covariates was successful. The gender, marital status, employment, nationality, and smoking behavior variables will be all tested at baseline using Chi-square to demonstrate that they are not significantly different between groups. Independent t-tests will be run at baseline measurements of dependent variables to make sure the study groups will be not significantly different on these variables before introducing the study intervention. One-way- ANOVA will be used to test the study hypotheses. Post hoc t-tests will be run to examine if the study groups will be significantly different on the dependent variables at end of the intervention. In case of having confounding effects of some variables, ANCOVA will be used.

Ethical consideration

Physical or psychological harm or risks that might be associated with the measurement activities or intervention employed in the current study will be minimal. One risk that might have resulted from the study was making venipuncture-related pain. Thus, ELMA cream has been used before blood sampling to decrease venipuncture-related pain. Moreover, trained nurses will draw blood from participants, following the Blood Sampling Guideline of the European Federation of Clinical Chemistry and Laboratory Medicine, 2017.

Potential benefits of the measurement activities and intervention to study subjects included increased knowledge and awareness about their health and mind-body modalities. For society, potential benefits included a greater understanding of the effects of mind-body modalities on stress reduction and the potential improvement of the study population's health. In this study, potential benefits are believed to exceed risks.

To protect the ethical principle of respect for subjects, all subjects will be informed about the purpose and nature of the study, and informed consent will be obtained from all. Students will be assured that they have the full right to refuse to participate in the study, and that such refusal will not affect their academic achievements in any way. They will also be assured that their information would not be made available to others without prior consent, the study data will be locked in a secured storage area in a locked locker and that their names will be replaced by numbers to avoid their identification. Also, the meetings with students will be conducted in a private room at JUST and at convenient times for subjects. Moreover, to meet the ethical principle of justice, no student will be excluded from the study because of gender, ethnicity, or nationality.

ELIGIBILITY:
Inclusion Criteria:

* Jordanian undergraduate nursing students
* Being 18 years old or older.
* Taking a clinical course.

Exclusion Criteria:

* Practicing any type of relaxation techniques, such as yoga, guided imagery, meditation, cognitive behavioral therapy.
* Taking hypnotics, sedatives, anxiolytic, anti-depressant, anti-inflammatory drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Executive Functioning | 6 weeks
  The Barkley Deficits in Executive Functioning Scale- Short form (BDEFS-SF) (Adult version) will be used to measure executive functions including self-organization, self-restraint, self-motivation, self-regulation of emotion, and self-management to time. It is a self-reported scale consisting of 20 items measured using a 4-point Likert-type scale, ranging from Never or rarely (1) to Sometimes (2), Often (3), and Very often (4). The BDEFS-SF internal consistency was reported at an alpha of .92 in adult population. A confirmatory factor analysis supported the 5-factor structure of BDEFS in college students.
Depression | 6 weeks
  Depression will be measured by the General Health Questionnaire-9 (PHQ-9). It is reliable self-administered tool to evaluate the frequency of depressive symptoms in nursing students. It includes 9 items measured on a 4 likert scale (0= not at all, 3= nearly every day). The scores ranges from 0 to 27, with the higher scores indicated higher levels of depression.
Anxiety | 6 weeks
  Anxiety will be measured using the Greneral Health Questionnaire-7 (PHQ-7). It is a valid and reliable self-report questionnaire for assessing the frequency of symptoms of anxiety in nursing students. It includes 7 items measured on 4-point likert scale that ranges from 0 (not at all) to 3 (nearly every day0. The scores range from 0 to 21, with higher the total score indicates higher levels of anxiety.
Physical symptoms | 6 weeks
  The Patient Health Questionnaire -15 (PHQ-15) is a self-reported somatic symptoms subscale, derived from the full Patient-Health-Questionnaire. It is a 15-item instrument that assesses 15 common somatic symptoms. Subjects are asked to rate the severity of symptoms as 0 ("not bothered at all"), 1 ("bothered a little"), or 2 ("bothered a lot"). The score ranges from 0 to 30 and scores of ≥5, ≥10, ≥15 represent mild, moderate and severe levels of somatization respectively. Evidence supports reliability and validity of the PHQ-15 as a measure of physical symptoms in the general population.
Biomarkers | 6 weeks
  The procedure and protocol of ELISA will be followed to measure the concentrations of the neurotransmitters and hormones in plasma that include cortisol, C-reactive protein, Interleukins, melatonin, and leptin.
  Similar units of measurement will be used.

SECONDARY OUTCOMES:
Negative Emotions | 6 weeks
  The negative emotions will be measured by the Depression, Anxiety and Stress Scale - 21 (DASS-21). It includes 3 self-administered subscales developed to assess the negative emotional states of depression, anxiety and stress. The total scores for each subscale ranges from 0 to 42, with higher scores indicating more depression, anxiety and stress.
Mindfulness | 6 weeks
  Mindful Attention Awareness Scale (MAAS) will be used to measure dispositional mindfulness. It is one-dimensional scale including 15 items measured on a six-point Likert type scale, ranging from 1 (almost always) to 6 (almost never). The score range is between 15 and 90, with higher score indicting higher levels of mindfulness. The scale has shown strong psychometric properties when validated in college students. It showed acceptable level of reliability and validity in university students.
Perceived stress | 6 weeks
  The Perceived Stress Scale (PSS) is used to measure the degree to which situations in one's life are appraised as stressful (unpredictable, uncontrollable, and overloaded). It include 10 items measured on a 5-point Likert scale (0=never, 4= very often), which are relatively free of content specific to any subpopulation group. The scores range from 0 to 40 with higher score indicating higher levels of perceived stress. PSS has been validated for use with college students.
Coping behaviors | 6 weeks
  Nursing students' self-directed coping behaviors will be assessed by the Coping Behaviors Inventory (CBI). The CBI is used to identify nursing students' coping behaviors. It includes nineteen 5-point Likert-type items divided into four factors: avoidance behavior (efforts to avoid a stressful situation), 6 items; problem-solving behavior (efforts to manage or change the stress arising out of a stressful situation), 6 items; optimistic coping behavior (efforts to keep a positive attitude toward the stressful situation), 4 items; and transference behavior (efforts to transfer one's attention from the stressful situation to other things), 3 items. Higher scores for each factor indicate more frequent use and greater effectiveness of a certain type of coping behavior. It showed an acceptable levels of reliability and validity in nursing students.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pulido-Martos M, Augusto-Landa JM, Lopez-Zafra E. Sources of stress in nursing students: a systematic review of quantitative studies. International Nursing Review. 2012 Mar;59(1):15-25.
- [Background] Shaban IA, Khater WA, Akhu-Zaheya LM. Undergraduate nursing students' stress sources and coping behaviours during their initial period of clinical training: a Jordanian perspective. Nurse Educ Pract. 2012 Jul;12(4):204-9. doi: 10.1016/j.nepr.2012.01.005. Epub 2012 Jan 26. PMID 22281123
- [Background] Wolf L, Stidham AW, Ross R. Predictors of stress and coping strategies of US accelerated vs. generic Baccalaureate Nursing students: an embedded mixed methods study. Nurse Educ Today. 2015 Jan;35(1):201-5. doi: 10.1016/j.nedt.2014.07.005. Epub 2014 Aug 2. PMID 25127928
- [Background] Chan CK, So WK, Fong DY. Hong Kong baccalaureate nursing students' stress and their coping strategies in clinical practice. J Prof Nurs. 2009 Sep-Oct;25(5):307-13. doi: 10.1016/j.profnurs.2009.01.018. PMID 19751936
- [Background] Evans W, Kelly B. Pre-registration diploma student nurse stress and coping measures. Nurse Educ Today. 2004 Aug;24(6):473-82. doi: 10.1016/j.nedt.2004.05.004. PMID 15312957
- [Background] Kinlein SA, Karatsoreos IN. The hypothalamic-pituitary-adrenal axis as a substrate for stress resilience: Interactions with the circadian clock. Front Neuroendocrinol. 2020 Jan;56:100819. doi: 10.1016/j.yfrne.2019.100819. Epub 2019 Dec 19. PMID 31863788
- [Background] Knight EL, Jiang Y, Rodriguez-Stanley J, Almeida DM, Engeland CG, Zilioli S. Perceived stress is linked to heightened biomarkers of inflammation via diurnal cortisol in a national sample of adults. Brain Behav Immun. 2021 Mar;93:206-213. doi: 10.1016/j.bbi.2021.01.015. Epub 2021 Jan 28. PMID 33515741
- [Background] Markozannes G, Koutsioumpa C, Cividini S, Monori G, Tsilidis KK, Kretsavos N, Theodoratou E, Gill D, Ioannidis JP, Tzoulaki I. Global assessment of C-reactive protein and health-related outcomes: an umbrella review of evidence from observational studies and Mendelian randomization studies. Eur J Epidemiol. 2021 Jan;36(1):11-36. doi: 10.1007/s10654-020-00681-w. Epub 2020 Sep 25. PMID 32978716
- [Background] Shields GS, Sazma MA, Yonelinas AP. The effects of acute stress on core executive functions: A meta-analysis and comparison with cortisol. Neurosci Biobehav Rev. 2016 Sep;68:651-668. doi: 10.1016/j.neubiorev.2016.06.038. Epub 2016 Jun 28. PMID 27371161
- [Background] Higginbotham, H. (2013). A psychoeducational approach to improving college student mental health. (Electronic Thesis or Dissertation).
- [Background] Smith JC. Relaxation, meditation, & mindfulness: A mental health practitioner's guide to new and traditional approaches. Springer Publishing Company; 2005 Mar 4.
- [Background] Gillani NB, Smith JC. Zen meditation and ABC relaxation theory: an exploration of relaxation states, beliefs, dispositions, and motivations. J Clin Psychol. 2001 Jun;57(6):839-46. doi: 10.1002/jclp.1053. PMID 11344469
- [Background] Prato CA, Yucha CB. Biofeedback-assisted relaxation training to decrease test anxiety in nursing students. Nurs Educ Perspect. 2013 Mar-Apr;34(2):76-81. doi: 10.5480/1536-5026-34.2.76. PMID 23763019
- [Background] Matsumoto M, Smith JC. Progressive muscle relaxation, breathing exercises, and ABC relaxation theory. J Clin Psychol. 2001 Dec;57(12):1551-7. doi: 10.1002/jclp.1117. PMID 11745596
- [Background] Barkley RA. Barkley deficits in executive functioning scale (BDEFS). Guilford Press; 2011 Feb 1.
- [Background] Coffman TP. The psychometric properties of the Barkley Deficits in Executive Functioning Scale (BDEFS) in a college student population (Doctoral dissertation). The Florida State University, 2014.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Ren L, Wang Y, Wu L, Wei Z, Cui LB, Wei X, Hu X, Peng J, Jin Y, Li F, Yang Q, Liu X. Network structure of depression and anxiety symptoms in Chinese female nursing students. BMC Psychiatry. 2021 May 31;21(1):279. doi: 10.1186/s12888-021-03276-1. PMID 34059013
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Rathnayake S, Ekanayaka J. Depression, anxiety, and stress among undergraduate nursing students in a public university in Sri Lanka. International Journal of Caring Sciences. 2016 Sep 1;9(3):1020-32.
- [Background] Kocalevent RD, Hinz A, Brahler E. Standardization of a screening instrument (PHQ-15) for somatization syndromes in the general population. BMC Psychiatry. 2013 Mar 20;13:91. doi: 10.1186/1471-244X-13-91. PMID 23514436
- [Background] Westermann J, Hubl W, Kaiser N, Salewski L. Simple, rapid and sensitive determination of epinephrine and norepinephrine in urine and plasma by non-competitive enzyme immunoassay, compared with HPLC method. Clin Lab. 2002;48(1-2):61-71. PMID 11833678
- [Background] Sheu S, Lin HS, Hwang SL. Perceived stress and physio-psycho-social status of nursing students during their initial period of clinical practice: the effect of coping behaviors. Int J Nurs Stud. 2002 Feb;39(2):165-75. doi: 10.1016/s0020-7489(01)00016-5. PMID 11755447
- [Background] Kwekkeboom KL, Wanta B, Bumpus M. Individual difference variables and the effects of progressive muscle relaxation and analgesic imagery interventions on cancer pain. J Pain Symptom Manage. 2008 Dec;36(6):604-15. doi: 10.1016/j.jpainsymman.2007.12.011. Epub 2008 May 27. PMID 18504089

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05172804/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05172804/ICF_001.pdf